CLINICAL TRIAL: NCT05972213
Title: Phenotypic and Functional Characterization of Neutrophils and Eosinophils in Severe Asthma Treated With Biotherapy
Acronym: CaPHe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230345
Record Dates: First submitted 2023-07-04; First posted 2023-08-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: severe asthma; biotherapies
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 ml of serum
  1ml of plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Longitudinal group: 25 patients anticipated. Patients with :
  * Uncontrolled asthma: ACT score < 20 and/or at least one exacerbation in the last 6 months
  * Naïve biotherapy
  * Indication for initiation of biotherapy according to the referring pulmonologist (omalizumab, mepolizumab, benralizumab, dupilumab)
- Cross-sectional group: 80 patients anticipated.
  * Patient on biotherapy (omalizumab, mepolizumab, benralizumab, dupilumab) for at least 6 months.
  * Controlled asthma (ACT > 20 and no exacerbation for 6 months) or uncontrolled asthma (ACT < 20 and/or at least 1 exacerbation for 6 months).

SUMMARY:
Neutrophils and eosinophils can have different functions. Depending on their environment, they can be more or less active, with more or less inflammatory activity.

Biotherapies can reduce the number of inflammatory cells in the blood and bronchi. However, it is not known whether they have the ability to modify the functions of the remaining cells.

The aim of this study is to better understand the functioning of eosinophilic and neutrophil polynuclear drugs involved in the response to biotherapies in severe asthma. The hypothesis is that biotherapies modify the inflammatory functions of polynuclear cells, which would contribute to the effect of the drug on asthma.

DETAILED DESCRIPTION:
Between 3 and 10% of adult asthmatics have a severe form of the disease. The pathophysiology of asthma is dominated by chronic bronchial inflammation of type "T2"" with eosinophil infiltration whose role in bronchial reshuffling, hyperresponsiveness and maintenance of inflammation has been well documented. They are specifically targeted by monoclonal antibodies to IL (inter leukin)-5, IL-5R and IL-4/13.

There is a population of severe asthmatics called "non-T2" characterized by Th17 inflammation, production of IL-6, IL-8, IL-11, GM-CSF (Granulocyte-macrophage colony-stimulating factor) and IL-17 and preponderant bronchial recruitment of neutrophils, resulting in greater clinical severity and decreased sensitivity to corticosteroids. Neutrophils, not specifically targeted by the current therapies used, release reactive forms of oxygen, proteases, neutrophil extracellular traps (NETs) contributing to airway inflammation. The phenotypic heterogeneity, functional heterogeneity and plasticity of neutrophils has been studied in other pathologies but not specifically in asthma.

The response to biotherapies is not always optimal with a significant number of failures or escapes in clinical practice.

There are limited data on these eosinophilic and neutrophil leukocyte subpopulations in asthma, including phenotypic changes under biotherapies. Cellular functions have not been studied under treatment and clinical response is unknown. In addition, neutrophils and eosinophils are most often studied separately, while both cell types contribute to inflammation and can regulate each other.

This study hypothesize an impact of severe asthma biotherapies on the subpopulations and functionality of polynuclear drugs, contributing to the observed therapeutic effect.

This work could lead to a better understanding of the mechanisms of response to biotherapies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ Age < 85 years
* Severe asthma as defined by ERS/ATS (European Respiratory Society/American Thoracic Society) 2014: asthma requiring high doses of ICS (inhaled corticosteroid) combined with another control therapy (such as long-acting bronchodilators), whether or not patients are controlled

Longitudinal group:

* Uncontrolled asthma: ACT score < 20 and/or at least one exacerbation in the last 6 months
* Naïve about biotherapy
* Indication for the initiation of biotherapy according to the referring pulmonologist (omalizumab, mepolizumab, benralizumab, dupilumab)

Cross-sectional group:

* Patient on biotherapy (omalizumab, mepolizumab, benralizumab, dupilumab) for at least 6 months.
* Controlled asthma (ACT > 20 and no exacerbation for 6 months) or uncontrolled asthma (ACT < 20 and/or at least 1 exacerbation for 6 months).

Exclusion Criteria:

* Refusal to participate or opposition to data processing
* Patient under guardianship or with curators
* Patient on immunosuppressant (other than corticosteroids)
* Treatment with biotherapy for another indication
* Patient not affiliated to a social security scheme or state medical aid

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe asthmatic patients followed in the Pneumology A department at Bichat Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-04-21 (Estimated); Study Completion 2024-05-21 (Estimated)

PRIMARY OUTCOMES:
Measurement of the difference between the studied parameters of polynuclear cells measured at 6 months compared to those measured at the start of biotherapy. | 3 months for the longitudinal group and 9 months for the cross-sectional group
  The main objective will be to characterize the longitudinal evolution of markers measured at 6 months after initiation of biotherapy.
  These parameters will be studied on a fresh blood sample collected peripherally on a 7 mL EDTA (Ethylenediaminetetraacetic acid) tube and 5 mL dry tube on the day of inclusion at the time of day hospital or pulmonology consultation, before initiation and during a follow-up pneumology consultation/day hospital at 6 months post-initiation.

SECONDARY OUTCOMES:
Measure the level of asthma control 6 months after the start of treatment, defined by the ACT score | 3 months for the longitudinal group and 9 months for the cross-sectional group
  Secondary objectives will be to measure an association of markers
Measure the number of exacerbations in the previous 6 months | 3 months for the longitudinal group and 9 months for the cross-sectional group
  Secondary objectives will be to measure an association of markers
Measure the type of biotherapy used | 3 months for the longitudinal group and 9 months for the cross-sectional group
  Secondary objectives will be to measure an association of markers

CONTACTS AND LOCATIONS:
Overall Officials: Camille Taillé, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No